CLINICAL TRIAL: NCT01642979
Title: Phase II Study of the Levamisole Combined With Cyclosporine A in Patients With Classic Paroxysmal Nocturnal Hemoglobinuria
Brief Title: Safety and Efficacy of Levamisole Combined With Cyclosporine A in Patients With Classic Paroxysmal Nocturnal Hemoglobinuria
Acronym: PNH-2012
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Yizhou Zheng, Vice director of the therapeutic centre of anemic diseases, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PNH-2012
Record Dates: First submitted 2012-07-14; First posted 2012-07-17 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria; Hemoglobinuria; Hemoglobinuria, Paroxysmal; Proteinuria; Urination Disorders; Thrombosis; Bone Marrow Failure; Aplastic Anemia,; Anemia, Hemolytic
Keywords: Paroxysmal Nocturnal Hemoglobinuria; Anemia; Hematologic Diseases; bone marrow failure; Immunologic Factors; Physiological Effects of Drugs; Levamisole; cyclosporine A
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Hemoglobinuria; Proteinuria; Urination Disorders; Thrombosis; Bone Marrow Failure Disorders; Anemia, Aplastic; Anemia, Hemolytic; Anemia; Hematologic Diseases | interventions — Levamisole; Cyclosporine; Glucocorticoids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Levamisole+cyclosporin A+Glucocorticoids (Experimental): Levamisole+cyclosporin A+Glucocorticoids
  Interventions: Drug: Levamisole+cyclosporin A+Glucocorticoids
- cyclosporin A+Glucocorticoids (Active Comparator): cyclosporin A+Glucocorticoids
  Interventions: Drug: cyclosporin A+Glucocorticoids
- Glucocorticoids (Active Comparator): Glucocorticoids
  Interventions: Drug: Glucocorticoids

INTERVENTIONS:
Drug: Levamisole+cyclosporin A+Glucocorticoids — Levamisole 2.5mg/kg every other day cyclosporin A 1.5-2.5mg/kg every other day Glucocorticoids0.5-1mg/kg every day(prednisone)
  Other Names: Levamisole; cyclosporin A; Glucocorticoids
  Arms: Levamisole+cyclosporin A+Glucocorticoids
Drug: cyclosporin A+Glucocorticoids — cyclosporin A 1.5-2.5mg/kg every day Glucocorticoids0.5-1mg/kg every day(prednisone)
  Other Names: cyclosporin A; Glucocorticoids
  Arms: cyclosporin A+Glucocorticoids
Drug: Glucocorticoids — Glucocorticoids 0.5-1mg/kg every day(prednisone)
  Arms: Glucocorticoids

SUMMARY:
Paroxysmal nocturnal hemoglobinuria is an acquired chronic hemolytic anemia,this study is designed to evaluate the safety and efficacy of Levamisole combined with cyclosporine A in patients with classic paroxysmal nocturnal hemoglobinuria.

DETAILED DESCRIPTION:
Paroxysmal nocturnal hemoglobinuria (PNH) is an acquired clonal disorder of the hematopoietic stem cell characterized by intravascular hemolysis, hemoglobinuria, anemia, and thrombosis, Patients may be at high risk of thrombosis and may develop bone marrow failure or aplastic anemia, with low white blood cell and platelet counts,because the manifestation and pathologic processes are complicate,the treatment is very difficult,this study is designed to evaluate the safety and efficacy of Levamisole combined with cyclosporine A in patients with classic paroxysmal nocturnal hemoglobinuria

ELIGIBILITY:
Inclusion Criteria:

1. Clinical and biochemical signs of classic Paroxysmal Nocturnal Hemoglobinuria
2. Diagnosis confirmed by Ham's test or Flow cytometry Patients have any Flow cytometry data
3. patient should complete levamisole study for at least half a year

Exclusion Criteria:

1. Active infection which requires antibiotic treatment
2. Pregnant or lactating women
3. Epilepsy and mental illness
4. Kidney and liver function abnormal
5. patient who terminate ealy from levamisole study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients in each group in complete or partial remission | 6 months
  she got blood transfusion-independent,the hemoglobin became higher

SECONDARY OUTCOMES:
Side effects | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: yizhou zheng, doctor, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital,, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Background] Parker C, Omine M, Richards S, Nishimura J, Bessler M, Ware R, Hillmen P, Luzzatto L, Young N, Kinoshita T, Rosse W, Socie G; International PNH Interest Group. Diagnosis and management of paroxysmal nocturnal hemoglobinuria. Blood. 2005 Dec 1;106(12):3699-709. doi: 10.1182/blood-2005-04-1717. Epub 2005 Jul 28. No abstract available. PMID 16051736
- See also: CBD — http://www.chinablood.com.cn